CLINICAL TRIAL: NCT03295838
Title: Symptom, Alexithymia and Self-image Outcomes of Mentalization-Based Treatment for Borderline Personality Disorder: a Naturalistic Study
Brief Title: Outcomes of Mentalization-Based Treatment for Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Viktor Kaldo, Med PhD, clinical psychologist, associate professor, research team leader, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNR 2011/1909-31/3
Record Dates: First submitted 2017-09-14; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline personality disorder; Psychotherapy; Treatment outcome; Pragmatic clinical trials as topic; Mentalization-based treatment; Alexithymia
MeSH Terms: conditions — Borderline Personality Disorder; Affective Symptoms | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Intervention Model Description: Patients were selected using a research protocol with defined criteria, all patients that were intended to treat in the Mentalization-based Treatment program were followed over 18 months and assessed for primary and secondary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mentalization-based Treatment (Experimental): MBT was conducted according to the treatment manual developed by Bateman & Fonagy. Patients were offered individual sessions with a psychotherapist and group sessions with 6-8 participants and 1-2 group therapists for 18 months. An introductory psycho-educational component (9-12 sessions) was also offered focusing on explicit mentalising skills (i.e. understanding one's own or others' intentions). Group and individual MBT focused on implicit mentalising towards self and others.
  Interventions: Behavioral: Mentalization-based treatment

INTERVENTIONS:
Behavioral: Mentalization-based treatment — See Arm description

SUMMARY:
The effects of a psychological treatment, Mentalization-Based Treatment, was studied using a research protocol with patients with mood swings and impulsive behavior (borderline personality disorder).

DETAILED DESCRIPTION:
Background: Mentalization-based treatment (MBT) in borderline personality disorder (BPD) has a growing evidence base, but there is a lack of effectiveness and moderator studies. The present study examined the effectiveness of MBT in a naturalistic setting and explored psychiatric and psychological moderators of outcome. Method: Borderline and general psychiatric symptoms, suicidality, self-harm, alexithymia and self-image were measured in a group of BPD patients (n=75) receiving MBT; assessments were made at baseline, and subsequently after 6, 12 and 18 months (when treatment ended). Borderline symptoms were the primary outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* To be included, BPD diagnosis was confirmed by SCID-II interview and the Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) interview, together with a consensus discussion between MBT therapists using DSM-IV and ICD-10 criteria. All patients referred between 2007-02-01 and 2012-05-30 were eligible for inclusion.

Exclusion Criteria:

* Exclusion criteria were: IQ<85, psychotic disorder other than schizotypal personality disorder, acute/temporary psychosis, previously diagnosed autism-spectrum disorder, bipolar disorder type I and severe eating or substance use disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identification.
Enrollment: 75 (Actual)
Dates: Start 2007-02-01 (Actual); Primary Completion 2014-05-03 (Actual); Study Completion 2014-05-03 (Actual)

PRIMARY OUTCOMES:
Borderline Symptoms | 0-18 months
  Key psychiatric and borderline symptomatology as measured by the Karolinska Borderline And Symptoms Scales (KABOSS-S) was the primary outcome measure. The KABOSS-S consists of three general symptom scales (depression, anxiety, obsessive-compulsive symptoms) derived from the Comprehensive Psychopathological Self-rating Scale for Affective Syndromes and one specific borderline scale compromising the items "Mood swings", "Ability to understand own emotions", "Self-control", "Self-soothing", "Feelings of abandonment", "Feelings of emptiness", "Self-image" and "Reality Presence". Each item is scored on a Likert scale from 0 ("no presence") to 6 ("severe").

SECONDARY OUTCOMES:
Suicidality | 0-18 months
  Suicidality was measured by the Suicide Assessment Scale, Self-Report (SUAS-S), which covers factors known to influence suicide risk, such as affect, bodily states, control and coping, emotional reactivity, as well as suicidal thoughts and behaviour.
General Psychiatric Symptoms | 0-18 months
  General psychiatric symptoms were measured using the Symptom Checklist-90 Revised (SCL-90-R), an established instrument with well-known reliability and validity.
Self-harm | 0-18 months
  Self-harm was measured by the Deliberate Self-Harm Inventory-9 (DSHI-9), which has well-known reliability and validity. This measure was introduced halfway through the study period (N=42).
Alexithymia | 0-18 months
  The Toronto Alexithymia Scale-20 (TAS-20) was used to measure alexithymia. It comprises 20 items divided into three subscales: Difficulty Identifying Feelings, Difficulty Expressing Feelings and Externally Oriented Thinking. TAS-20 was used to measure affective mentalization.
Self-image | 0-18 months
  Self-image was assessed using Structural Analysis of Social Behavior (SASB). SASB is based on a circumplex model, measuring self-image and interpersonal interactions in relation to three interpersonal "surfaces" (i.e. actions of others, reactions to others and the introject, or what can be called the self-image. The third surface (self-image) was used, which comprises eight clusters of self-image: 1) Autonomy; 2) Self-affirmation; 3) Active self-love; 4) Self-protection; 5) Self-control; 6) Self-blame; 7) Self-attack; and 8) Self-neglect.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Yes
The dataset used and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 1st feb 2007 - 3rd may 2014.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Derived] Lof J, Clinton D, Kaldo V, Ryden G. Symptom, alexithymia and self-image outcomes of Mentalisation-based treatment for borderline personality disorder: a naturalistic study. BMC Psychiatry. 2018 Jun 11;18(1):185. doi: 10.1186/s12888-018-1699-6. PMID 29890960